CLINICAL TRIAL: NCT01734005
Title: Efficacy and Safety of Red Ginseng on Decrement of Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ARIMED-BF-GC
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Ginseng (Experimental)
  Interventions: Dietary Supplement: Red Ginseng
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Red Ginseng — Red Ginseng (1.4g/day)
  Arms: Red Ginseng
Dietary Supplement: Placebo — Placebo (1.4g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of red ginseng on decrement of body fat. The investigators measured decrement of body fat parameters , including Body Fat Mass, Percent Body Fat, weight and BMI(body mass index), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-65 years old
* BMI(body mass index) ≥ 25 kg/m^2 or WC(Waist Circumference) ≥ 90(men), WC ≥ 85(women)
* Able to give informed consent

Exclusion Criteria:

* Significant variation in weight(more 10%) in the past 3 months
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in Body Fat Mass | 12 weeks
  Body Fat Mass was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Percent Body Fat | 12 weeks
  Percent Body Fat was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in weight | 12 weeks
  Weight was measured in study visit 1(0 week) and visit 3(12 week).
Changes in BMI(body mass index) | 12 weeks
  BMI(body mass index) was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea